CLINICAL TRIAL: NCT06634498
Title: The Effect of Repetitive Transcranial Magnetic Stimulation of the Left Dorsolateral Prefrontal Cortex in Internet Gaming Disorder
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation for Internet Gaming Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jin-tao Zhang (Other)
Collaborators: Zi-Liang Wang, Medical Ethics Committee of Zhenjiang Mental Health Center (Unknown)
Responsible Party: Sponsor-Investigator, Jin-tao Zhang, Professor, Beijing Normal University
Organization: Beijing Normal University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: The effect of rTMS in IGD
Record Dates: First submitted 2024-10-05; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Internet Gaming Disorder
Keywords: rTMS; Internet gaming disorder; craving; craving regulation
MeSH Terms: conditions — Internet Addiction Disorder | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: within-subject, sham-controlled design: all subjects will receive active and sham rTMS in a randomized order
Who Masked: Participant, Investigator
Masking Description: single blind: both participants and experiment won't know the stimulation condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real rTMS on the dlPFC (Experimental): rTMS on the DLPFC Dorsolateral prefrontal cortex (DLPFC) target will be identified by the baseline functional magnetic resonance imaging (fMRI) study for regulation of craving using a separate sample. During the intervention, each participant will receive an iTBS mode intervention on this DLPFC region.
  Interventions: Other: real rTMS on the dlPFC
- sham rTMS on the dlPFC (Sham Comparator): Each participant will also receive a sham rTMS intervention as a controlled condition.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: real rTMS on the dlPFC — During real rTM session, participants will perform the regulation of craving (ROC). In the rest phase, participants need to relax and rest. In the ROC task, participants will regulate craving elicited by gaming pictures using cognitive reappraisal. During the task, reaction times (RTs) and craving scores wil be recorded.
  Arms: real rTMS on the dlPFC
Other: Sham (No Treatment) — During the sham rTMS session, participants will perform the regulation of craving (ROC). In the ROC task, participants will regulate craving elicited by gaming pictures using cognitive reappraisal. During the task, reaction times (RTs) and craving scores wil be recorded.
  Arms: sham rTMS on the dlPFC

SUMMARY:
This study aims to investigate the intervention effects of navigated repetitive transcranial magnetic stimulation (rTMS) on craving regulation in individuals with internet gaming disorder (IGD). The primary objectives include: (1) examining the impact of navigated rTMS over the dorsolateral prefrontal cortex (DLPFC) on the gaming cravings, and craving regulation capacity; and (2) exploring the potential neural mechanisms by which rTMS over the DLPFC improves craving intensity, and craving regulation ability.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) has been shown to reduce cravings in individuals with substance addiction. However, to date, no studies have systematically examined the short-term and long-term clinical and cognitive effects of sustained rTMS treatment on internet gaming disorder (IGD). This study seeks to fill that gap by adopting a within-subject design to investigate the cognitive (craving regulation capacity) and neural (structural changes, resting-state and task-related brain activity, and functional connectivity between the dorsolateral prefrontal cortex [DLPFC] and reward-related brain regions) effects of personalized and precisely navigated rTMS treatment in individuals with IGD.

Participants will receive both real intermittent theta-burst stimulation (iTBS) and sham stimulation targeting the left DLPFC. The study aims to assess how these interventions influence clinical and neural outcomes. Specifically, the experiment will measure changes in craving regulation capacity, and neural markers including resting-state functional connectivity and task-evoked activation patterns in key brain regions associated with addiction, such as the DLPFC and reward system.

The entire experimental protocol spans three weeks and follows a randomized crossover design. Participants will be randomly assigned to one of two intervention sequences: real iTBS followed by sham stimulation, or sham stimulation followed by real iTBS. Each rTMS session will utilize iTBS parameters, lasting approximately 10 minutes, with a minimum of one week between the two sessions to avoid potential carryover effects.

To evaluate the effects of the interventions, clinical assessments (Craving scores), cognitive measures (craving regulation ability), and neuroimaging data (fMRI at rest and during task performance) will be collected after each intervention session. This approach allows for a comprehensive assessment of both the short-term and potential cumulative effects of rTMS on cognitive and neural correlates of IGD, contributing valuable insights into the mechanisms by which rTMS may modulate addictive behaviors and associated neural circuits.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V gaming disorder >5 and scored ≥ 50 on a revised version of Young's online Internet addiction test；
* spent more than 50% of their online time gaming；
* engagement in one of four popular Internet game (Arena of Valor,Genshine, LOL, FPS) for over 20 hours per week for at least 1 year.

Exclusion Criteria:

* current or history of use of illegal substances and gambling;
* current or history of psychiatric or neurological illness;
* current use of psychotropic medications;
* cognitive impairment as assessed by the Mini-International Neuropsychiatric Interview；
* surgery, head trauma or heart related diseases in the past year；
* a history of epilepsy or seizures or increased risk of seizures for any reason；
* metal implants or tattoos of the neck or head；
* claustrophobia.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in craving scores in the Cue-Reactivity(CR) task | Approximately 10 minutes during real rTMS condition and sham rTMS
  Comparing the participants who reported craving scores for the game stimuli in the unregulated condition and in the regulated condition in the CR task conducted separately during real rTMS and sham rTMS. Higher scores mean higher craving.
Changes in the DLPFC and craving-related brains (striatum, amygdala) activities in the ROC task following rTMS and sham rTMS | Approximately 14 minutes - 29 minutes after real rTMS and sham rTMS
  This study will compare the changes in DLPFC activity during the ROC task after real rTMS and sham rTMS. In addition, craving-related brain regions (striatum and amygdala) are also concerned.
Alterations in the functional connectivity between the DLPFC and other brain regions in the ROC task following rTMS and sham rTMS | Approximately 14 minutes - 29 minutes after real rTMS and sham rTMS
  The present study compares the alterations in functional connectivity between the DLPFC and other brain regions (especially those related to reward) after real TMS and sham TMS.

SECONDARY OUTCOMES:
Changes in ReHo and fALFF/ALFF in resting-state following rTMS and sham rTMS | 5 minutes-13 minutes after real rTMS and sham rTMS
  This study will compare changes in brain regional homogeneity (ReHo) and the fractional amplitude of low-frequency fluctuations (fALFF/ALFF) during the resting state following real rTMS and sham rTMS, particularly in the DLPFC and reward-related brain regions. These measures reflect the effects of rTMS on participants.
The DLPFC-based functional connectivity alterations during resting-state fMRI | 5 minutes-13 minutes after real rTMS and sham rTMS
  Use seed -based functional connectivity method to explore the alterations in the functional connectivity between the DLPFC and other brain regions, particularly reward-related areas, will be examined.
The intra- and inter-connectivity within brain networks during resting-state fMRI | 5 minutes-13 minutes after real rTMS and sham rTMS
  Graph-theoretic analysis will be used to depict alterations in brain networks following real rTMS and sham rTMS. The present study also concern the changes in intra- and inter-connectivity within brain networks (including executive control systems, reward systems, and default networks) after real rTMS and sham rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tao Zhang, Phd, Principal Investigator — Beijing Normal University
Locations (2):
- China (2):
  - Medical Ethics Committee of Zhenjiang Mental Health Center, Zhenjiang, Jiangsu
  - State Key Laboratory of Cognitive Neuroscience and Learning, Beijing

IPD SHARING:
Plan to Share IPD: Undecided